CLINICAL TRIAL: NCT00871754
Title: Molecular Analysis Of Bladder Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Lahey Clinic (Other)
Responsible Party: Principal Investigator, Linda Topjian, study coordinator, Lahey Clinic
Other Study IDs: 88-009A
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer; Bladder Neoplasms
Keywords: Bladder Cancer; Cancer, bladder; Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a laboratory study where the investigators hope to look at chromosomal events implicated in bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient's undergoing removal of a malignant bladder tumor
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 1988-04; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Reiger-Christ, PhD, Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States